CLINICAL TRIAL: NCT04161729
Title: Effects of Intraoperative Magnesium Sulfate on Pain Relief, Hemodynamics and Quality of Recovery After Spine Surgery
Brief Title: Effects of Intraoperative Magnesium Sulfate on Perioperative Pain Relief After Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Georgia Tsaousi, Assistant Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SpiMag
Record Dates: First submitted 2019-11-03; First posted 2019-11-13 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Analgesia; Pain, Postoperative; Spine Disease
Keywords: magnesium; analgesia; pain score; opioid consumption; spine surgery
MeSH Terms: conditions — Agnosia; Pain, Postoperative; Spinal Diseases | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium sulfate (Active Comparator): Magnesium sulfate 20 mg/kg intravenous over a 15-min period before induction of anesthesia and 20 mg/kg/h by continuous i.v. infusion until surgery completion.
  Interventions: Drug: Magnesium Sulfate; Drug: Isotonic saline 0.9%
- Isotonic solution 0.9% (Placebo Comparator): Isotonic solution 0.9% in the same volume as the study drug using identical pattern of administration.
  Interventions: Drug: Magnesium Sulfate; Drug: Isotonic saline 0.9%

INTERVENTIONS:
Drug: Magnesium Sulfate — Intravenous magnesium sulfate 20 mg/kg in 100ml isotonic saline 0.9% over a 15-min period before induction of anesthesia and 20 mg/kg/h by continuous i.v. infusion until surgery completion.
Drug: Isotonic saline 0.9% — Isotonic saline 0.9% 100ml over a 15-min period before induction of anesthesia and thereafter continuous i.v. infusion until surgery completion in dosage identical to magnesium sulfate group.

SUMMARY:
The treatment of postoperative pain is increasingly based on a multimodal approach and although opioids remain the drug of choice, they are often used in combination with other analgesics (paracetamol, cyclooxygenase inhibitors or non-steroidal anti-inflammatory drugs) and co-analgesic agents (clonidine and anti- NMDA such as ketamine or MgSO4). The rationale for combined analgesia is to achieve additive or synergistic analgesic properties while decreasing the incidence of side effects by reducing the dose of each agent. Nociceptive stimuli are known to activate the release of the excitatory amino acid glutamate in the dorsal horn of the spinal cord. The resultant activation of NMDA receptors causes calcium entry into the cell and triggers central sensitisation. This mechanism is involved in the perception of pain and mainly accounts for its persistence during the postoperative period.

Although magnesium is not a primary analgesic in itself, it enhances the analgesic actions of more established analgesics as an adjuvant agent. Magnesium produces a voltage-dependent block of NMDA receptors and has been reported to have analgesic properties that might be related to this inhibiting property. Magnesium sulfate has been reported to be effective in perioperative pain treatment and in blunting somatic, autonomic and endocrine reflexes provoked by noxious stimuli.

When magnesium was used intraoperatively, many researchers reported that it reduced the requirement for anesthetics and/or muscle relaxants.

Intraoperative use of magnesium sulfate can also be associated with decreased incidences of nausea and vomiting after surgery, which could have been due to the lower consumption of anesthetics (i.e. volatile agents), rather than any antiemetic effect of magnesium sulfate. In addition, perioperative i.v. administration of magnesium sulfate has another advantageous effect, as it decreases the incidence of shivering by up to 70-90%. Previous studies investigating the analgesic efficacy of MgSO4 in general, gynaecological, ophthalmic and orthopaedic surgery have shown conflicting results, while reports regarding spine surgery are extremely limited.

Our study was designed to investigate the effects of MgSO4 on perioperative pain relief and postoperative quality of recovery after lumbar laminectomy surgery.

DETAILED DESCRIPTION:
Each participant will receive standard monitoring (ECG, SpO2, capnography, SBP, oesophageal temperature, accelerography) and an intravenous access will be established. The level of anaesthesia will be monitored with the bispectral index (BIS), targeting to a BIS level 40-50.

Group M patients will receive intravenous magnesium sulfate 20 mg/kg over a 15-min period before induction of anaesthesia and 20 mg/kg/h by continuous i.v. infusion during the operation. Group C will be given isotonic solution of 0.9% in the same volume as the study drug.

A standard anesthesia protocol will be applied involving propofol 2mg/kg (iv) and fendanyl 2 μg/kg (iv). Cis-atracurium 0.2 mg/kg (iv) will be given to facilitate endotracheal intubation. Anaesthesia will be maintained with air 50% and oxygen 50%, and desflurane adjusted to achieve a target BIS between 40 and 50. Remifentanil will be added to the anesthesia regimen as needed.

Hemodynamic parameters will be recorded upon

* Baseline: Before the administration of the tested drug
* T5: 5 minutes after the administration of the tested drug
* T10: 10 minutes after the administration of the tested drug
* T15: 15 minutes after the administration of the tested drug
* Ts: surgical incision
* T30: 30 minutes after the administration of the tested drug
* T45: 45 minutes after the administration of the tested drug
* T60: 60 minutes after the administration of the tested drug
* T90: 90 minutes after the administration of the tested drug
* T120: 120 minutes after the administration of the tested drug
* T180: 180 minutes after the administration of the tested drug

Low arterial blood pressure during surgery defined as a mean blood pressure value < 50 mmHg will be treated by a bolus of 5 mg ephedrine administered intravenously or phenylephirne civ for persistent hypotension.

Also, time to accelerography recording indicating the appropriateness of neuromuscular block for intubation, mean expired desflurane concentration (from 30 min after skin incision to the end of surgery), boluses of ephedrine and total intraoperative remifentanil consumption will be recorded.

Postoperative analgesic protocol will involve paracetamol 1 mg (iv), lornoxicam 8mg (iv) and morphine 3 mg (upon request).

Postoperatively pain assessment will be performed by Visual Analogue Scale (VAS), Verbal Rating Scale (VRS) and Numerical Rating Scale (NRS) at emergence from anesthesia and 2, 4, 6, and 24 h in the study period. Time to first analgesic request and total analgesics consumption postoperatively (morphine equivalents) will be recorded. Episodes of shivering, as well as episodes of nausea and vomiting (PONV), will be recorded at emergence and thereafter, throughout the study period. Finally, patients' global satisfaction will be assessed the first day after surgery using a 5-grade scale (1= worst discomfort ever experienced in their life and 5= totally satisfied during the immediate postoperative period).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 18 and 80 years
* ASA Physical status 1 to 3
* Elective or semi-elective lumbar laminectomy surgery
* Signed informed consent

Exclusion Criteria:

* Under medication with calcium channel blockers or magnesium
* Drugs or alcohol abuse
* Neurological disorders
* Myopathy
* Intracardiac block
* Hepatic failure
* Renal failure
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-05-03 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Analgesics consumption postoperatively in morphine equivalents | 24 hours after the emergence from anesthesia
  The difference in analgesic consumption (assessed as mg of morphine equivalents) postoperatively after intravenous infusion of magnesium sulfate or isotonic saline 0.9%

SECONDARY OUTCOMES:
Analgesics consumption intraoperatively | 180 minutes intraoperatively
  The difference in analgesics consumption (μg of remifentanil) intraoperatively after /during intravenous infusion of magnesium sulfate or isotonic saline 0.9%
Pain intensity | 10 minutes after emergence from anesthesia, 2, 4 and 6 hours after the emergence from anesthesia
  The difference in pain intensity postoperatively assessed by Visual Analogue Scale, Numerical Pain Scale or Verbal Pain Scale after intravenous infusion of magnesium sulfate or isotonic saline 0.9%
Time to first analgesic request in minutes | 24 hours after the emergence from anesthesia
  The difference in the time frame (minutes) for analgesia request after emergence from anesthesia after intravenous infusion of magnesium sulfate or isotonic saline 0.9%

OTHER OUTCOMES:
Heart rate changes intraoperatively | 180 minutes intraoperatively
  The changes in heart rate (beats per minute) intraoperatively after /during intravenous infusion of magnesium sulfate or isotonic saline 0.9%
Systemic blood pressure changes intraoperatively | 180 minutes intraoperatively
  The changes in systemic blood pressure (mmHg) intraoperatively after /during intravenous infusion of magnesium sulfate or isotonic saline 0.9%
Postoperative adverse effects | 24 hours after the emergence from anesthesia
  The incidence of shivering and nausea /vomiting after emergence from anesthesia after intravenous infusion of magnesium sulfate or isotonic saline 0.9%
Patients' satisfaction | 24 hours after surgery
  The patients' global satisfaction assessed the day after surgery using a 5-grade scale (1= worst and 5= totally satisfied) after intravenous infusion of magnesium sulfate or isotonic saline 0.9%

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Tsaousi, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No